CLINICAL TRIAL: NCT05764044
Title: Adjuvant Chemotherapy in Cell-free Human Papillomavirus Deoxyribonucleic Acid (cfHPV-DNA) Plasma Positive Patients: A Biomarker In Locally Advanced Cervical Cancer (CC)
Brief Title: Adjuvant Chemotherapy in cfHPV-DNA Plasma Positive Patients: A Biomarker In Locally Advanced Cervical Cancer
Acronym: AddChemo
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AddChemo CC Trial
Record Dates: First submitted 2023-03-01; First posted 2023-03-10 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer; Cervix Cancer; Cervix Neoplasm
Keywords: Human papillomavirus; HPV; Cervical cancer; Circulating free DNA; Adjuvant chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, multicenter, national, superiority, parallel, clinical trial, design to evaluate the use of adjuvant chemotherapy in patients with locally advanced cervical cancer, selected by cfDNA-HPV biomarker. Intervention arm will count on application of two additional cycles of cisplatin-based adjuvant chemotherapy 50mg/m2 D1 and gemcitabine 1000mg/m2 D1 and D8 at every 21 days. Randomization will be allocated 1:1. Participants will be followed at every 4 months, in person or by phone. Primary endpoint is progression-free survival time.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Standard of Care) (Other): Patients will be followed with plasma cfDNA-HPV, computed tomography (CT) scan of the thorax and magnetic resonance (MRI) of abdomen and pelvis and clinical and gynecological examination at every four months.
  Interventions: Other: Follow-up
- Experimental Arm (Experimental): Receive two cycles of cisplatin-based adjuvant chemotherapy 50mg/m2 D1 and gemcitabine 1000mg/m2 D1 and D8 at every 21 days. After that, patients will be followed with plasma cfDNA-HPV, computed tomography (CT) scan of the thorax and magnetic resonance (MRI) of abdomen and pelvis and clinical and gynecological examination at every four months.
  Interventions: Drug: cisplatin, gemcitabine; Other: Follow-up

INTERVENTIONS:
Drug: cisplatin, gemcitabine — Two additional cycles of cisplatin-based adjuvant chemotherapy 50mg/m2 D1 and gemcitabine 1000mg/m2 D1 and D8 at every 21 days.
  Arms: Experimental Arm
Other: Follow-up — Patients will be followed with plasma cfDNA-HPV, computed tomography (CT) scan of the thorax and magnetic resonance (MRI) of abdomen and pelvis and clinical and gynecological examination at every four months.

SUMMARY:
This study hypothesizes that patients who persist with cell-free human papillomavirus deoxyribonucleic acid (cfHPV-DNA) plasma expression at the end of standard treatment, can derive the benefit of using adjuvant chemotherapy in locally advanced cervical cancer (CC). After standard treatment based on concomitant chemoradiotherapy regime, a qualitative and quantitative research of cfHPV-DNA in plasma of patients will be conducted. Patients who have positive research for plasma cfHPV-DNA at the end of chemoradiotherapy treatment will be randomized to receive two additional cycles of adjuvant chemotherapy or observation. Patients will be followed with conduction of computed tomography (CT) scan of the thorax and magnetic resonance (MRI) of abdomen and pelvis and clinical and gynecological examination at every four months.

DETAILED DESCRIPTION:
A prospective, randomized, multicenter, national, superiority, parallel, clinical trial, design to evaluate the use of adjuvant chemotherapy in patients with locally advanced cervical cancer selected by cfDNA-HPV biomarker. Patients will be randomized by stratified randomization process to belong to one of the groups: control (Group B) or intervention (Group C), emphasizing homogeneity of risk factors between them. A randomized list will be generated by using a suitable software, using variable size blocks (2 or 4), with stratification for site and staging. The confidentiality of the randomization list will be maintained through an automated, centralized, Internet-based randomization system, available 24 hours a day (RedCap). Selected patients must receive standard treatment based on concomitant chemoradiotherapy regime, with dose of radiation of 40-50 greys (Gy) (considering additional boost of 10-15 Gy in lymph nodes, radiologically or surgically, compromised) and brachytherapy of 30-40 Gy and cisplatin 40mg/m2 weekly. After four weeks of the end of treatment, a qualitative and quantitative research of cfHPV-DNA in plasma of patients will be conducted. Those with a negative qualitative research result will leave the study. Patients who have positive research for plasma 16, 18, 26, 31, 33, 35, 39, 45, 51, 52, 53, 56, 58, 59, 66, 68, 69, 73, 82 cfHPV-DNA at the end of chemoradiotherapy treatment will be randomized to receive two additional cycles of adjuvant chemotherapy or observation. In those cases in which the duration of radiochemotherapy treatment exceeds 84 days, patients must undergo imaging examination (chest, abdomen and pelvis CT) in order to exclude pre-randomization metastatic disease. Patients will be followed with conduction of computed tomography (CT) scan of the thorax and magnetic resonance (MRI) of abdomen and pelvis and clinical and gynecological examination at every four months.

ELIGIBILITY:
Inclusion Criteria:

* International Federation of Gynecology and Obstetrics (FIGO) 2018 stage IB3 to IVA will be included prospectively.
* Previous standard treatment based on concomitant chemoradiotherapy regimen.
* Karnofsky performance status score ≥70, with estimated life expectancy ≥12 weeks,
* Immunocompetent,
* Positive research for types 16, 18, 26, 31, 33, 35, 39, 45, 51, 52, 53, 56, 58, 59, 66, 68, 69, 73, 82 cfHPV-DNA in plasma at the end of chemoradiotherapy,
* Proper hematological, liver and kidney functions. Inclusion criteria will include absolute neutrophils count ≥1.5 x 109/L, platelets ≥100 x 10/L, serum bilirubin ≤ 2.0 x upper limit of normal (ULN), calculated creatinine clearance ≥50 mL/min and alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase ≤ 2.5 x ULN.
* Patients of child-bearing potential were obligated to use an approved contraceptive method during and for 3 months after the study;
* Agree with research procedures, by signing the Informed Consent Form (ICF).

Exclusion Criteria:

* Previous cervical cancer or other malignancies,
* Pregnant women,
* Inability to perform concurrent cisplatin based-chemoradiotherapy.
* Tumors containing different HPV genotypes
* Absence of anatomopathological examination to prove the diagnosis and/or staging examinations.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 120 days
  Progression-free survival will be calculated from the date of randomization until the date of progression, whether local or distant, or death.

SECONDARY OUTCOMES:
Overall survival | 120 days
  Pverall survival will be calculated from the date of randomization until death or last follow-up. Follow-up will be updated at each consultation and the following possibilities will be considered: living without disease, living with disease, death from cancer, death from another cause and loss of follow-up.
Overall response rate | 120 days
  Response assessment will be performed using RECIST 1.1 (2009) criteria through pelvic MRI. Thus, complete response (CR) will be considered the disappearance of all lesions. Partial response (PR), reduction (30%) in the sum of the largest diameters of target lesions, when compared to the initial examination. Disease progression (PD): increase (20%) in the sum of the largest diameters of the lesions, when compared to the initial examination or the appearance of new lesions. Stable disease: does not meet criteria for PR or PD.
Quality of life measures (EORTC QLQ-C30 and QLC-CX24) | 21 to 120 days
  Generic quality of life measures (EORTC QLQ-C30) will be assessed during medical consultations in this clinical study, considering that this questionnaire alone does not adequately assess specific treatment issues that affect the quality of life of women with cervical cancer, a QLQ-CX24 add-on module will also be applied. All questionnaires used in this study are self-administered, however, in those cases where the ability to understand, little education/illiteracy is considered low or when telephone monitoring is in force, the tests will be applied by the researchers, who will seek to read all the questions and help mark answers.
Toxicity according to the Common Terminology Criteria for Adverse Events v.5.0 | 7 to 120 days
  Toxicity will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (2017). Hematological (anemia, neutropenia, thrombocytopenia and febrile neutropenia), gastrointestinal (diarrhea, nausea and vomiting), renal (serum creatinine changes) and hepatic (AST and ALT changes) toxicities will be evaluated. Grade 1 and 2 toxicities, together, were considered mild and grade 3 and 4 toxicities were considered severe.

CONTACTS AND LOCATIONS:
Locations (26):
- Brazil (26):
  - Centro Integrado de Pesquisa da Amazônia, CINPAM, Manaus, Amazonas
  - Hospital Evangélico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital Samur, Vitória da Conquista, Estado de Bahia
  - Hospital de Base do Distrito Federal, Brasília, Federal District
  - Hospital do Câncer de Muriaé, Muriaé, Minas Gerais
  - Centro de Oncologia de Cascavel, CEONC, Cascavel, Paraná
  - União Oeste Paranaense de Estudos e Combate ao Câncer, UOPECCAN, Cascavel, Paraná
  - Centro Integrado de Oncologia de Curitiba, CIONC, Curitiba, Paraná
  - Instituto Nacional do Câncer, INCA, Rio de Janeiro, Rio de Janeiro
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Hospital Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Hospital Geral de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Centro Gaúcho Integrado Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Centro Oncologico de Roraima, CECOR, Boa Vista, Roraima
  - Catarina Pesquisa Clínica, Itajaí, Santa Catarina
  - Hospital Unimed, Joinville, Santa Catarina
  - Centro de Atenção Integral a Saúde da Mulher, CAISM, Campinas, São Paulo
  - Hospital do Amor, Jales, São Paulo
  - Hospital da Mulher - SECONCI, São Paulo, São Paulo
  - Hospital do Coração - Research Institute, São Paulo, São Paulo
  - Instituto Brasileiro de Combate ao Câncer, IBCC São Camilo, São Paulo, São Paulo
  - Hospital São Paulo, Unifesp, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Centro de Estudos e Pesquisa de Hematologia, CEPHO, São Paulo, São Paulo
  - Instituo de Câncer Brasil, ICB, Taubaté, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Data could be shared after reasonable request of the principal investigator.
Supporting Information: Study Protocol
Time Frame: After study completion.